CLINICAL TRIAL: NCT00090415
Title: UW STAART Center of Excellence
Brief Title: Early Characteristics of Autism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U54MH066399 (NIH); U54MH066399 (NIH); DDTR BD-DD
Record Dates: First submitted 2004-08-26; First posted 2004-08-27 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Autism; Autistic Disorder
Keywords: Autism; Developmental Delay Disorders
MeSH Terms: conditions — Autistic Disorder; Developmental Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Child participants with autism will undergo intensive behavioral therapy.
  Interventions: Behavioral: Intensive behavioral therapy
- 2 (No Intervention): Child participants without autism will receive no treatment and will undergo assessments to determine brain functioning only.

INTERVENTIONS:
Behavioral: Intensive behavioral therapy — Participants will undergo a magnetic resonance imaging (MRI) scan and will complete various activities to determine brain functioning. In addition, children with autism will take part in intensive behavioral therapy at least 4 hours every day for the duration of the study.
  Arms: 1

SUMMARY:
This study will identify factors that distinguish children with autism from children with developmental delay and those with normal development and study the efficacy of intensive behavioral therapy in children with autism.

DETAILED DESCRIPTION:
Children with autism often suffer from social, educational, and functional problems. By understanding the social, linguistic, psychological, and physiological differences that distinguish between autistic children, developmentally delayed children, and children with typical development, researchers may be able to recognize autism early in life so that children with autism can be helped as early as possible and their long-term outcome can be improved.

Children in this study will be enrolled for 2 years. They will receive annual evaluations throughout the two-year period. They will undergo a magnetic resonance imaging (MRI) scan and will complete various activities to determine brain functioning. In addition, children with autism will take part in intensive behavioral therapy at least 4 hours every day for the duration of the study. Communication and social behavior scales, an early development interview, observations of parent/child interaction, and neuropsychological, cognitive, and adaptive behavioral measures will be used to assess participants.

ELIGIBILITY:
Inclusion Criteria for Autistic Participants:

* Diagnosis of autism

Inclusion Criteria for Developmentally Delayed Participants:

* Exhibiting current delays in development

Inclusion Criteria for Participants with Normal Development:

* Exhibiting normal development

Inclusion Criteria for All Participants:

* Overall good health

Ages: 18 Months to 30 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2003-04; Primary Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Communication and social behavior scales; an early development interview; observations of parent/child interaction; and neuropsychological, cognitive, and adaptive behavioral measures | Measured at Year 2

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Aylward, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Dawson G, Rogers S, Munson J, Smith M, Winter J, Greenson J, Donaldson A, Varley J. Randomized, controlled trial of an intervention for toddlers with autism: the Early Start Denver Model. Pediatrics. 2010 Jan;125(1):e17-23. doi: 10.1542/peds.2009-0958. Epub 2009 Nov 30. PMID 19948568